CLINICAL TRIAL: NCT02504424
Title: AirXpanders AeroForm Tissue Expander System for Breast Reconstruction (XPAND-II)
Brief Title: AirXpanders AeroForm Tissue Expander System for Breast Reconstruction
Acronym: XPAND-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AirXpanders, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP-0005 AirXpanders
Record Dates: First submitted 2015-07-20; First posted 2015-07-22 (Estimated); Results first posted 2018-09-05 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2019-01

CONDITIONS: Breast Cancer
Keywords: Tissue Expansion; Tissue Expander; Breast Tissue Expansion; Breast Tissue Expander; Breast Reconstruction; 2 Stage Breast Reconstruction
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AeroForm Tissue Expander (Experimental): AeroForm Tissue Expansion inflation with carbon dioxide by remote control
  Interventions: Device: AeroForm Tissue Expander

INTERVENTIONS:
Device: AeroForm Tissue Expander — The AeroForm Tissue Expander is a breast tissue expander implanted following mastectomy and activated by remote control to release small doses of carbon dioxide from an internal reservoir to fill and inflate the expander.

SUMMARY:
This study is designed to allow existing investigators continued access to the AeroForm Tissue Expander to treat patients while AirXpanders completes a marketing application and during the review process by FDA.

DETAILED DESCRIPTION:
This is a prospective, multi-center, single arm, open-label, continued access clinical study. Subjects who meet the inclusion criteria and agree to participate in the study will be enrolled and implanted with the investigational AeroForm Tissue Expander. If the subject is having a bilateral procedure, the AeroForm expander will be implanted in each side. Subjects will be followed until the first post-operative visit after explant of the tissue expander(s) and exchange for permanent implant(s).

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between the ages of 18-70
* Subject requires tissue expansion as part of breast reconstruction
* Subject is able to provide written informed consent
* Subject is able and willing to comply with all of the study requirements
* Subject has the physical, perceptual and cognitive capacity to understand and manage the at home dosing regimen

Exclusion Criteria:

* Subject's tissue integrity is unsuitable for tissue expansion
* Subject has residual gross malignancy at the intended expansion site
* Subject has current or prior infection at the intended expansion site
* Subject has a history of failed tissue expansion or breast reconstruction
* Subject has any co-morbid condition determined by the Investigator to place the subject at an increased risk of complications (e.g., severe collagen vascular disease, poorly managed diabetes)
* Subject is taking any concomitant medications determined by the Investigator to place the subject at an increased risk of complications (e.g., Prednisone, Coumadin).

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2015-11-12 (Actual); Primary Completion 2017-05-03 (Actual); Study Completion 2017-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Jacobs, M.D., Study Chair — AirXpanders Chief Medical Officer; Jeffrey Ascherman, M.D., Principal Investigator — Columbia University
Locations (8):
- United States (8):
  - Marin General Hospital, Greenbrae, California
  - Good Samaritan Hospital, San Jose, San Jose, California
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Faulkner Hospital, Boston, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - Columbia University, New York, New York
  - Presbyterian Medical Center, Charlotte, North Carolina

REFERENCES:
- [Derived] Ascherman JA, Zeidler K, Morrison KA, Appel J, Castle J, Chun Y, Colwell A, Mohebali K, Stokes T, Sudarsky L. Results of XPAND II: A Multicenter, Prospective, Continued-Access Clinical Trial Using the AeroForm Tissue Expander for Two-Stage Breast Reconstruction. Plast Reconstr Surg. 2020 Jan;145(1):21e-29e. doi: 10.1097/PRS.0000000000006395. PMID 31881599

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited women who were planning to have immediate or delayed breast reconstruction (unilateral or bilateral) post-mastectomy and required tissue expansion to develop tissue coverage for placement of standard breast implant(s). Subjects were identified from the medical practice of the participating investigators.
Groups:
- AeroForm Tissue Expander: AeroForm Tissue Expansion inflation with carbon dioxide gas by remote control
  AeroForm Tissue Expander: The AeroForm Tissue Expander is a breast tissue expander implanted following mastectomy and activated by remote control to release small doses of carbon dioxide gas from an internal reservoir to fill and inflate the expander.
Period: Overall Study
Arm/Group | AeroForm Tissue Expander
Started | 50
Completed | 48
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: 50 Subjects treated under protocol
Groups:
- AeroForm Tissue Expander: AeroForm Tissue Expansion inflation with carbon dioxide gas by remote control
  AeroForm Tissue Expander: The AeroForm Tissue Expander is a breast tissue expander implanted following mastectomy and activated by remote control to release small doses of carbon dioxide from an internal reservoir to fill and inflate the expander.
Arm/Group | AeroForm Tissue Expander
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 47
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 42
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 40
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 50
Body Mass Index [Mean (Standard Deviation); unit: lbs/in^2] | 24.5 (3.57)

OUTCOME MEASURES:

1. Primary Outcome: Number of Breasts With Successful Tissue Expansion With Exchange to a Permanent Breast Implant Unless Exchange is Precluded by a Non-device Related Event
Description: The primary endpoint is analyzed per breast. Breasts in which the expander is removed and/or replaced due to a device related adverse event or a device malfunction are counted as failures.
Time Frame: 6 months
Population: * of participants is 48: # treated (50) minus participant failed exchange of both breasts for non-device related reason (1) and participant not analyzed due to withdrawal (1).
  * of breasts is 80: # breasts treated (86) minus # breasts failed exchanged due to non-device related reason (4) and # breasts not analyzable due to withdrawal (2).
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | AeroForm Tissue Expander
Number analyzed (Participants) | 48
Number analyzed (breasts) | 80
breasts | 80
Statistical Analysis 1: Comparison: AeroForm Tissue Expander; Treatment Success includes all breasts which were exchanged successfully in the Per Protocol Cohort, excluding non-device related failures. The Treatment Success Rate per breast is 100% (80/80). Note: Denominator = 80 (86 implanted breasts - 6 breasts). Failed exchange = 4 breasts (non-device related) & Missing = 2 breasts (patient non-compliant w/study and withdrew consent after treatment); Test type: Other; percent of breasts successfully exchange = 100
Statistical Analysis 2: Comparison: AeroForm Tissue Expander; Sensitivity Analysis (Best / Worst Case): Treatment Success by subject for the Per Protocol cohort includes all failures (excluding non-device related failures). The best case analysis considers success if the subject has at least one breast successfully reconstructed, and the worst case analysis considers it a failure if at least one breast has failed. The treatment success by subject is 100% for both best and worst case analysis; Test type: Other; % breasts successfully exchanged = 100

2. Secondary Outcome: Number of Breast With Successful Tissue Expansion With Exchange to Permanent Implant Including All Breasts in the Per Protocol Cohort.
Description: Secondary analysis is repeated including all breasts in the PP cohort (including non-device related failures). The Treatment Success Rate by breast, based on the Per Protocol cohort, including all cause failures, is 95.2% (80/84). One subject (2 breasts) are not included in the analyses due to not completing the second stage surgery and withdrawal of consent.
Time Frame: 6 months
Population: Analysis population includes all treated breasts with the exception of 2 breasts that were not exchanged at the time of study completion (subject withdrew from study)
Measure: Count of Units; unit: breasts
Units Other Than Participants: breasts
Arm/Group | AeroForm Tissue Expander
Number analyzed (Participants) | 49
Number analyzed (breasts) | 84
breasts | 80
Statistical Analysis 1: Comparison: AeroForm Tissue Expander; Secondary analysis is repeated including all breasts in the PP cohort (including non-device related failures). The Treatment Success Rate by breast, based on the Per Protocol cohort, including all cause failures, is 95.2% (80/84). One subject (2 breasts) are not included in analysis as subject withdrew from the study prior to exchange of her expanders; Test type: Other; % breasts successfully exchanged = 95.2

ADVERSE EVENTS:
Time Frame: 1 year
Description: The safety of the device is evaluated by:
  * Device related adverse events
  * All adverse events, regardless of whether serious or there is a causal relationship to the device.
  * Serious device related adverse events
  * All serious adverse events, regardless of whether there is a causal relationship to the device.
  * Device malfunctions leading to expander removal and/or replacement.
Arm/Group | AeroForm Tissue Expander
All-Cause Mortality (participants affected / at risk) | 0/50
Serious Adverse Events (participants affected / at risk) | 11/50
Other Adverse Events (participants affected / at risk) | 8/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroForm Tissue Expander (N=50)
cellulitis (Reproductive system and breast disorders) | 4 (4)
wound dehiscence (Reproductive system and breast disorders) | 1 (1)
hematoma (Reproductive system and breast disorders) | 1 (1)
seroma (Reproductive system and breast disorders) | 1 (1)
neutropenic fever, weakness (Immune system disorders) | 1 (1)
inflammation (red breast syndrome) (Reproductive system and breast disorders) | 2 (2)
urinary tract infection (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AeroForm Tissue Expander (N=50)
erythema (Skin and subcutaneous tissue disorders) | 5 (5)
seroma (Reproductive system and breast disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02504424/Prot_SAP_000.pdf